CLINICAL TRIAL: NCT07161557
Title: An Open Observational Study to Evaluate Metabolic Health in People Aged 18 to 60 by Nutrilite Metabolic Health Index
Brief Title: Evaluating Metabolic Health in People Aged 18 to 60 by Nutrilite Metabolic Health Index
Status: Not yet recruiting | Type: Observational
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-RD-10-AY-001
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Abnormality; Metabolic Disorders
Keywords: Diet2Me; Nutrilite Metabolic Health Index; Metabolic health omics model; Metabolomics testing
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants enrolled will be asked to fill out the questionnaires, have physical checkup, and take blood samples, no interventions involved.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention involved, participants will fill out some questionnaires and blood samples will drawn for test and analysis.

SUMMARY:
The goal of this observational study is to evaluate Metabolic Health by fit analysis between calculated Nutrilite Metabolic Health Index and the result of Metabolomics analysis from blood plasma samples in healthy adult participants aged between 18 and 60 years. The main question it aims to answer:

- Does the Nutrilite Metabolic Health Index fit well with the result of Metabolomics analysis from blood plasma samples?

200 eligible participants will be enrolled in a single center, one site visit will be made to finish a health questionnaire, a lifestyle questionnaire, a routine physical checkup. Blood samples will be collected for routine blood test (blood sugar, total triglycerides, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, uric acid), and for Metabolomics testing.

Researchers will calculate the Nutrilite Metabolic Health Index based on participant data, and do the fit analysis against the result from Metabolomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers, aged 18 to 60, regardless of gender;
* Not participating in other interventional clinical studies;
* Have a good understanding of the nature, purpose, benefits obtained, and possible risks and side effects of the study;
* Willing to comply with all trial requirements and procedures;
* Sign the informed consent form.

Exclusion Criteria:

* In the treatment of gastrointestinal symptoms;
* Those who are lactose intolerant, allergic to fish and their products;
* Current suffering from other organic diseases affecting bowel function, such as history of gastrointestinal resection, colon or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, Hirschsprung's disease, scleroderma, anorexia nervosa, etc.;
* Diet control, exercise enhancement, or taking medications that control weight or affect appetite in the past 3 months;
* Volunteers have any of the following medical history or have been clinically diagnosed with the following diseases that may affect the evaluation of the test results: obvious gastrointestinal disorders, liver, kidney, endocrine, blood, respiratory and cardiovascular diseases;
* Current or past abuse of alcohol or other illicit drugs, supplements, or OTC prescriptions 3 / 11 Research content Collection of biological samples or information data Evaluation indicators Drugs may cause intestinal dysfunction or affect the evaluation of trial effects;
* Frequent use of drugs that may affect gastrointestinal function or immune system according to the investigator's judgment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female participants, aged 18 to 60, regardless of gender;
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-09 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Nutrilite Metabolic Health Index | day 1
  Nutrilite Metabolic Health Index incorporates seven core biochemical parameters (see details in Secondary Outcome Measures): body mass index (BMI), waist circumference, fasting blood glucose (FBG) level, blood lipid profile (total cholesterol (TC), total triglycerides(TG), Low-Density Lipoprotein Cholesterol (LDL), High-Density Lipoprotein Cholesterol (HDL), blood pressure (Systolic Blood Pressure(SBP), and Diastolic Blood Pressure (BDP)), uric acid level, and history of fatty liver disease; along with four lifestyle and hereditary factors: smoking, alcohol consumption, age, and family history of metabolic diseases.
  After weighted calculation, the index score ranges from 0 to 100, divided into four grades:
  Excellent: 85-100 Moderate: 60-84 Poor: 40-59 Severe: 0-39

SECONDARY OUTCOMES:
SBP | day 1
  SBP(Systolic Blood Pressure), ideally <120 mmHg or still normal if less than 130mmHg
DBP | day 1
  BDP(Diastolic Blood Pressure), ideally <80 mmHg, or still normal if less than 89 mmHg
Blood test - LDL-C | day 1
  LDL-C(Low-Density Lipoprotein Cholesterol) concentration level in the blood sample test: normal range 0-3.1mmol/L, higher than 3.1 mmol/L is abnormal;
Blood test - HDL-C | day 1
  HDL-C(High-Density Lipoprotein Cholesterol) concentration level in the blood sample test: normal range 1.04~1.55 mmol/L, lower than 1.04 or higher than 1.55 mmol/L is abnormal;
Blood test - TG | day 1
  TG (Triglyceride) concentration level in the blood sample test : normal range 0~1.7 mmol/L, higher than 1.7mmol/L is abnormal
Blood test - TC | day 1
  TC (Total Cholesterol) concentration level in the blood sample test: normal range 3-5.2 mmol/L; higher than 5.2 mmol/L is abnormal.
Blood test - FBG | day 1
  FBG(Fasting Blood Glucose) concentration level in the blood sample test: normal range 4.-5.5mmol/L, higher than 5.5 mmol/L is abnormal.
BMI | day 1
  BMI (Body Mass Index), BMI is calculated by weight/height^2, where weight measured with unit kg, and height with unit meter, and weight and height will be combined to report BMI in kg/m^2.
Waist Circumference | day 1
  waist circumference measured in cm (centimeter)
Uric Acid Level | day 1
  uric acid level in μmol/L, the normal range for adult male：149～416μmol/L, adult female：89～357μmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Qu, Principal Investigator — Shanghai MCC Hospital
Locations (1):
- Shanghai MCC Hospital, Shanghai, Shanghai Municipality, China